CLINICAL TRIAL: NCT03983343
Title: Skin Glues Compared to Running Sutures for Perineal Skin Repair After Vaginal Delivery. A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0039-19-EMC
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Perineal Tear
Keywords: Adhesive glue; Episiotomy; Pain sensation; Perineal tears; Running sutures; Skin closure; Visual Analogue Scale

STUDY DESIGN:
Intervention Model Description: Eligible patients will be asked to participate in this trial before perineal tear repair.
  The patients will be randomly assigned to one of the two groups in a 1:1 ratio:
  1. Suturing the perineal skin of the perineum using fast-absorbable running sutures (Vicryl Rapide 3-0)
  2. Closing the perineal skin using adhesive glue- exofin® (Octyl-2-cyanoacrylate). Other than skin closure, both groups will be treated similarly according to standard protocol used for perineal tear repair. In both groups, the walls of the vagina, the perineal muscles and the subcutaneous tissue will be repaired and approximated using the standard method, i.e. with running sutures using Vicryl Rapid Stitch 2-0.
Who Masked: Outcomes Assessor
Masking Description: Cosmetic result will be assessed 4-6 weeks after the repair by a doctor who did not participate in tear suturing immediately after delivery, and is not aware to the repair method used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- control group (No Intervention): Standard technique: Suturing the perineal skin with fast-absorbable running sutures (Vicryl Rapide 3-0).
- intervention group (Active Comparator): Closing the perineal skin using adhesive glue- exofin® (Octyl-2-cyanoacrylate)
  Interventions: Device: exofin®

INTERVENTIONS:
Device: exofin® — Perineal skin will be closed by adhesive glue - exofin® (Octyl-2-cyanoacrylate).
  Arms: intervention group

SUMMARY:
The incidence of a perineal tears during labor is 70 to 90%, while in 96% of the cases it's a minor perineal tear (grade 1). In about 3% to 4% the perineal tear is major and involve the external (grade 3) and the internal anal sphincter (grade 4). Episiotomy, which is considered an iatrogenic grade 2 tear, is performed in about 12% of vaginal deliveries.

Complications related to perineal tears include bleeding, the most common, that may lead to the development of vaginal or perineal hematoma. Additionally, local infection can develop and complicate the recovery from the injury. In rare cases, abscesses may occur and in rarer cases necrotizing fasciitis or recto-vaginal fistula may also evolve.

The "gold standard" method for repairing perineal tears is to use absorbable (preferably fast-absorbing) sutures. Grade 1 tears that do not bleed and do not disrupt the anatomical structure of the perineum usually do not require repair. Grade 2 tears are usually sewn in a continuous absorbent suture and less in the form of single stitches.

The use of adhesive glue to repair skin injuries began 20 years ago and the main adhesive used is dermabond® (Ethicon Inc. octyl-2-cyanoacrylate). The use of glue is faster and lead to less pain than the use of stitches or staples. It can be used for a variety of large or small, traumatic or iatrogenic wounds, with a cosmetic result, infection rate, and dehiscence rate similar to those achieved by stitches or staples.

In light of this, the investigators intend to conduct a randomized trial that will examine the advantages and disadvantages of the use of glue compared to the traditional sutures for closure of the skin in perineal tears grade 1 and 2 and episiotomies after vaginal delivery.

The investigators hypothesis is that the use of adhesive glue to close the skin in perineal tears grade 1 and 2 (including episiotomy), will be faster and associated with less pain compared to the traditional suturing method, without a significant difference in the rate of complications.

DETAILED DESCRIPTION:
Trial design: Randomized controlled trial.

Objectives: To examine the effect of adhesive glue compared to fast-absorbable running sutures on pain sensation following repairing perineal skin in cases of tears grade 1 and 2.

Trial population: Women delivering vaginally at Emek Medical Center, and experience a spontaneous perineal tear, grade 1 or 2, or episiotomy.

Trial course:

Eligible patients will be asked to participate in this trial before perineal tear repair. Following providing an explanation about the trial, patients will be asked to provide written informed consent to participate in the trial.

The patients will be randomly assigned to one of the two groups in a 1:1 ratio:

1. Suturing the perineal skin of the perineum using fast-absorbable running sutures (Vicryl Rapide 3-0)
2. Closing the perineal skin using adhesive glue- exofin® (Octyl-2-cyanoacrylate). Other than skin closure, both groups will be treated similarly according to standard protocol used for perineal tear repair.

Sample size In order to detect a reduction of 20% in the VAS (visual analogue pain score) within 2 hours of the procedure between the groups [from 40% to 20% in the running sutures and glue groups, respectively) with a level of significance of 95% (α = 0.05 - two tailed) and a power of 80% (β = 0.2) a sample size of 182 women (91 per group) is needed.

Data collected during the study:

* Data collected during the repair of the tear: maternal age, ethnicity, pre-gestational body mass index, background medical conditions, medication use, smoking status, birth's number, number of vaginal/caesarean births in the past, perineal tears in the past, antenatal complications, gestational age at delivery, epidural use during labor, birth weight, gender, grade of tear, spontaneous or episiotomy, cross over (failure of completing the procedure with the assigned method), number of skin sutures/glue capsules that was used, length of the perineal incision, repair time, use of local analgesics during repair, pain sensation related to the procedure. Pain sensation will be evaluated within 2 hours using a 0 (no pain) to 100 Visual Analogue Scale (VAS). Additionally immediate breastfeeding will be assessed as well.
* Data collected 48 hours after the repair and prior to discharge: pain level during walking/standing/sitting/lying down, (pain will be evaluated using the same VAS), discomfort during walking/standing/sitting/lying down, difficulty and pain in urination, local edema, local infection, separation of the edges of the wound, need for re-suturing, need to remove a stitch, woman's satisfaction and breastfeeding.
* Data collected 4-6 weeks after repair: women will be asked to return for check-up visit by a physician that was not involved in the repair and unaware of the allocation group. The outcomes that will be assessed at this visit will include: pain during walking/standing/sitting/lying, discomfort during walking/standing/sitting/lying down, difficulty and pain in urination, time to return to sexual activity, dyspareunia, cosmetic result, skin dehiscence and granuloma, preference of women for the next delivery. A telephone questionnaire will be used to collect the same data among women who do not attend the clinic visit within 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-45.
2. Term birth (> 37.0 weeks).
3. Perineal tears grade 1 or 2, or episiotomy.

Exclusion Criteria:

1. Perineal tears grades 3 or 4.
2. Operative vaginal deliveries.
3. Significant background diseases that can affect pain or recovery time: Pregestational diabetes mellitus, any heart disease, severe pulmonary disease, collagen or connective tissue disease, rheumatic diseases, autoimmune diseases, known immunodeficiency and chronic steroid use.
4. Signs of local infection prior to the beginning of repair of the tear.
5. Known allergy to exofin®.
6. Pregestational body mass index > 35 kg/m2.
7. Women with excessive bleeding that does not allow the use of glue.
8. Delivery of a dead fetus.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 182 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | within 2 hours after completing the procedure
  Pain intensity will be measured by asking the woman to describe the pain related to the procedure using a 0 (no pain) to 100 VAS (intolerable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Emek Medical Center, Afula, Israel
Locations (1):
- EMEK Medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith LA, Price N, Simonite V, Burns EE. Incidence of and risk factors for perineal trauma: a prospective observational study. BMC Pregnancy Childbirth. 2013 Mar 7;13:59. doi: 10.1186/1471-2393-13-59. PMID 23497085
- [Background] Vale de Castro Monteiro M, Pereira GM, Aguiar RA, Azevedo RL, Correia-Junior MD, Reis ZS. Risk factors for severe obstetric perineal lacerations. Int Urogynecol J. 2016 Jan;27(1):61-7. doi: 10.1007/s00192-015-2795-5. Epub 2015 Jul 30. PMID 26224381
- [Background] Friedman AM, Ananth CV, Prendergast E, D'Alton ME, Wright JD. Variation in and factors associated with use of episiotomy. JAMA. 2015 Jan 13;313(2):197-9. doi: 10.1001/jama.2014.14774. No abstract available. PMID 25585333
- [Background] Kalis V, Laine K, de Leeuw JW, Ismail KM, Tincello DG. Classification of episiotomy: towards a standardisation of terminology. BJOG. 2012 Apr;119(5):522-6. doi: 10.1111/j.1471-0528.2011.03268.x. Epub 2012 Feb 3. PMID 22304364
- [Background] Leeman L, Rogers R, Borders N, Teaf D, Qualls C. The Effect of Perineal Lacerations on Pelvic Floor Function and Anatomy at 6 Months Postpartum in a Prospective Cohort of Nulliparous Women. Birth. 2016 Dec;43(4):293-302. doi: 10.1111/birt.12258. Epub 2016 Oct 31. PMID 27797099
- [Background] Kettle C, Dowswell T, Ismail KM. Continuous and interrupted suturing techniques for repair of episiotomy or second-degree tears. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD000947. doi: 10.1002/14651858.CD000947.pub3. PMID 23152204
- [Background] Feigenberg T, Maor-Sagie E, Zivi E, Abu-Dia M, Ben-Meir A, Sela HY, Ezra Y. Using adhesive glue to repair first degree perineal tears: a prospective randomized controlled trial. Biomed Res Int. 2014;2014:526590. doi: 10.1155/2014/526590. Epub 2014 Jun 26. PMID 25089271
- [Background] Singer AJ, Thode HC Jr. A review of the literature on octylcyanoacrylate tissue adhesive. Am J Surg. 2004 Feb;187(2):238-48. doi: 10.1016/j.amjsurg.2003.11.017. PMID 14769312
- [Background] Seijmonsbergen-Schermers AE, Sahami S, Lucas C, Jonge Ad. Nonsuturing or Skin Adhesives versus Suturing of the Perineal Skin After Childbirth: A Systematic Review. Birth. 2015 Jun;42(2):100-15. doi: 10.1111/birt.12166. Epub 2015 Apr 11. PMID 25864727
- [Background] Mota R, Costa F, Amaral A, Oliveira F, Santos CC, Ayres-De-Campos D. Skin adhesive versus subcuticular suture for perineal skin repair after episiotomy--a randomized controlled trial. Acta Obstet Gynecol Scand. 2009;88(6):660-6. doi: 10.1080/00016340902883133. PMID 19353332
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 198: Prevention and Management of Obstetric Lacerations at Vaginal Delivery. Obstet Gynecol. 2018 Sep;132(3):e87-e102. doi: 10.1097/AOG.0000000000002841. PMID 30134424
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 165: Prevention and Management of Obstetric Lacerations at Vaginal Delivery. Obstet Gynecol. 2016 Jul;128(1):e1-e15. doi: 10.1097/AOG.0000000000001523. PMID 27333357